CLINICAL TRIAL: NCT05000021
Title: Reducing Diabetes Distress Using Cognitive Behavioral Therapy in Young Adults With Type 1 Diabetes
Acronym: ReDUCe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); DexCom, Inc. (Industry); Breakthrough T1D (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-12789; 4-SRA-2021-1071-M-B (Other Grant/Funding Number: JUVENILE DIABETES RESEARCH FOUNDATION (JDRF))
Record Dates: First submitted 2021-07-26; First posted 2021-08-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; diabetes distress; young adult; cognitive behavioral therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Cognitive Behavioral Therapy; Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cognitive Behavioral Therapy for Diabetes Distress (CBT-DD) with Continuous Glucose Monitoring (Experimental): Participants randomized to this arm will receive Cognitive Behavioral Therapy for Diabetes Distress (CBT-DD), enhanced by review of Continuous Glucose Monitoring (CGM) data. Participants will wear study-supplied CGM for the first 6 months of their participation in the trial.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Diabetes Distress (CBT-DD) with Continuous Glucose Monitoring; Device: Continuous Glucose Monitoring (CGM)
- Continuous Glucose Monitoring (CGM) Only (Active Comparator): Participants randomized to receive Continuous Glucose Monitoring (CGM) will continue to receive their usual care and will also wear CGM throughout the first 6 months of their participation in the trial.
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Diabetes Distress (CBT-DD) with Continuous Glucose Monitoring — CBT-DD consists of approximately 10 individual sessions of CBT delivered virtually by trained protocol therapists, conducted over the course of approximately 12 weeks. The CBT-DD consists of 5 core modules targeting negative emotionality and aversive reactions to emotional experiences. These modules are preceded by an introductory session that reviews the patient's presenting symptoms and provides a therapeutic rationale, as well as a module on motivational enhancement. The final module consists of relapse prevention. CBT-DD sessions will integrate a review of Continuous Glucose Monitoring (CGM) data and feedback will be provided by the therapist.
  Arms: Cognitive Behavioral Therapy for Diabetes Distress (CBT-DD) with Continuous Glucose Monitoring
Device: Continuous Glucose Monitoring (CGM) — Use of commercially available, FDA-approved continuous glucose monitoring (CGM) for 6 months post-randomization. Usual diabetes care will continue and participants can initiate a CGM review from their healthcare providers, as desired. In addition, a nurse practitioner with expertise in CGM will train each participant via video recordings in the proper placement of the device, and technical issues, and provide basic teaching at the beginning of the trial on interpretation of CGM data and self-titration of insulin/self-management. Written materials and online resources for recognizing and managing diabetes distress, along with self-management information and treatment options to discuss with providers will also be provided.

SUMMARY:
This project proposes to use telemedicine-delivered cognitive-behavioral therapy (CBT) enhanced with continuous glucose monitor (CGM) review to target diabetes distress in adults with type 1 diabetes. The efficacy of CBT for diabetes distress (CBT-DD) will be tested in comparison to commercial FDA-approved CGM only in a randomized controlled clinical trial. The investigators' central hypothesis is that the addition of a CBT intervention that targets diabetes distress and self-management directly will yield clinically significant improvements in both diabetes distress and glycemic control relative to CGM alone. The investigators propose to recruit 93 adults (age 18-64) with type 1 diabetes from a national population for an entirely virtual 6-month study over four years, with targeted recruitment of racial/ethnic minorities. In addition to standard measurement of HbA1c for glycemic control and validated patient-reported outcome (PRO) surveys, the investigators plan to innovatively integrate momentary psychological and behavioral data via smartphone-based ecological momentary assessment with CGM data to assess day-to-day changes in diabetes distress, affect, self-management, and glycemia over the course of the trial.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial (RCT) of CBT-DD, enhanced by CGM feedback. The study period will last for 6 months, with the first 3 months on CGM and consisting of a 2-week run-in period prior to randomization, in which ecological momentary assessment (EMA) data will be collected daily, followed by an 8-week CBT intervention period in which EMA data will be collected weekly surrounding CBT sessions, with a subsequent 2-week period post-intervention in which EMA data will again be collected daily. Both intervention and control groups will be doing the same EMA and CGM procedures to enable matching data for comparison. Follow-up virtual study data collection will occur at 3, 6, 9, and 12 months to assess the primary outcome of HbA1c and durability of intervention effect on diabetes distress and HbA1c. Participants in both arms will be provided a sufficient supply of CGM sensors to track their blood glucose daily, throughout the first 6 months of the study. If participants already have personal CGM, they will replace with study-supplied CGM.

We will also collect qualitative information from people with Type 1 Diabetes (T1D) ages 35-64 to solicit suggestions and inform future study decisions. We will create 2-4 focus groups to ask their impressions about our current study and explore key factors like establishing adult care and attending medical appointments, disease self-management, and adjusting to chronic disease. We will compare interview responses from participant groups who have high vs. low social needs and poor vs. good glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes (T1D) duration ≥6 months
* English or Spanish speaking
* At least moderate Diabetes Distress (DD) (score of ≥2 on T1D-Diabetes Distress Scale)
* Stable insulin treatment regimen (insulin prescription, use of pump, etc.) for at least 3 months prior to study enrollment

Exclusion Criteria:

* Comorbid psychiatric condition, including depression, anxiety, or suicidality, which may be independently associated with the main outcomes of DD or glycemic control. Comorbid psychiatric conditions listed above are being excluded because CBT-DD currently centers on mitigating specifically diabetes distress to improve glycemic outcomes
* In treatment for a psychological condition within the last 6 months or on a non-stable dose of psychiatric medication over the last 2 months
* Developmental or sensory disability interfering with participation
* Current pregnancy, as self-management and glycemic goals differ
* Participation in another behavioral intervention study
* Use of non-insulin medications or recent medical procedures that would impact glycemic control or use of CGM over the study
* Minors
* Subjects who do have the capacity to consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress Levels | Baseline and 3 months post-intervention
  Diabetes distress will be assessed using the Problem Areas in Diabetes (PAID) scale. The PAID scale will be administered to each participant via the REDCap database. The PAID scale is a 20 item, self-report questionnaire that describes negative emotions related to diabetes commonly experienced by people with diabetes. For each item, participants are asked to provide a response describing the extent the item is currently a diabetes issue for them using a 5-point Likert scale ranging from 0 ("Not a problem") to 4 ("Serious problem"). Scores are added and multiplied by 1.25, yielding an overall possible score of 0-100. Scores will be summarized by study arm using basic descriptive statistics. Patients scoring >=40 may be at the level of "emotional burnout" and warrant special attention.

SECONDARY OUTCOMES:
Hemoglobin A1c | 3 months post-intervention
  Hemoglobin A1c (HbA1c) values will be calculated using mailed point-of-care (POC) kits for home collection. Samples will be collected, returned, processed, and shipped for analysis by a central laboratory. HbA1c results will be summarized by study arm using basic descriptive statistics.
Time in Range (TIR) calculated from Continuous Glucose Monitoring (CGM) | Every 14 days through the first 3 months post-intervention
  The percentage of time glucose values were within range (i.e., between 70-180 mg/dL) will be calculated from CGM data during the 3 months after randomization. Results will be summarized by study arm using basic descriptive statistics.
Time Below Range (TBR) calculated from CGM | Every 14 days through the first 3 months post-intervention
  The percentage of time that glucose values were below range (i.e., ≤ 70 mg/dL and ≤ 55 mg/dL) will be calculated from CGM data during the 3 months after randomization. Percentage of TBR will be calculated for both thresholds. Results will be summarized by study arm using basic descriptive statistics.
Time Above Range (TAR) calculated from CGM | Every 14 days through the first 3 months post-intervention
  The percentage of time glucose values were above range (≥ 180 mg/dL and ≥ 250 mg/dL) will be calculated from CGM wear data during the 3 months after randomization. Percentage of TAR will be calculated for both thresholds. Results will be summarized by study arm using basic descriptive statistics.
Coefficient of Variation (CV) for Glycemic Variability | Every 14 days through the first 3 months post-intervention
  The CV for glycemic variability will be calculated based on the values obtained from CGM. CV, which is a measure of variability, is defined as the standard deviation of glucose changes divided by the mean glucose value and will expressed as a percentage. Results will be summarized by study arm.

OTHER OUTCOMES:
Diabetes Distress Levels | Baseline and 6 months, 9 months and 12 months post-intervention
  Diabetes distress will be assessed using the Problem Areas in Diabetes (PAID) scale. The PAID scale will be administered to each participant via the REDCap database. The PAID scale is a 20 item, self-report questionnaire that describes negative emotions related to diabetes commonly experienced by people with diabetes. For each item, participants are asked to provide a response describing the extent the item is currently a diabetes issue for them using a 5-point Likert scale ranging from 0 ("Not a problem") to 4 ("Serious problem"). Scores are added and multiplied by 1.25, yielding an overall possible score of 0-100. Scores will be summarized by study arm using basic descriptive statistics. Patients scoring >=40 may be at the level of "emotional burnout" and warrant special attention.
Hemoglobin A1c | 6 months, 9 months, and 12 months post-intervention
  Hemoglobin A1c (HbA1c) values will be calculated from mailed kits for home collection and analysis by a central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gonzalez, PhD, Principal Investigator — Yeshiva University
Locations (2):
- United States (2):
  - Yeshiva University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young-Hyman D, de Groot M, Hill-Briggs F, Gonzalez JS, Hood K, Peyrot M. Psychosocial Care for People With Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Dec;39(12):2126-2140. doi: 10.2337/dc16-2053. No abstract available. PMID 27879358
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Peters A, Laffel L; American Diabetes Association Transitions Working Group. Diabetes care for emerging adults: recommendations for transition from pediatric to adult diabetes care systems: a position statement of the American Diabetes Association, with representation by the American College of Osteopathic Family Physicians, the American Academy of Pediatrics, the American Association of Clinical Endocrinologists, the American Osteopathic Association, the Centers for Disease Control and Prevention, Children with Diabetes, The Endocrine Society, the International Society for Pediatric and Adolescent Diabetes, Juvenile Diabetes Research Foundation International, the National Diabetes Education Program, and the Pediatric Endocrine Society (formerly Lawson Wilkins Pediatric Endocrine Society). Diabetes Care. 2011 Nov;34(11):2477-85. doi: 10.2337/dc11-1723. No abstract available. PMID 22025785
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Livingstone SJ, Levin D, Looker HC, Lindsay RS, Wild SH, Joss N, Leese G, Leslie P, McCrimmon RJ, Metcalfe W, McKnight JA, Morris AD, Pearson DW, Petrie JR, Philip S, Sattar NA, Traynor JP, Colhoun HM; Scottish Diabetes Research Network epidemiology group; Scottish Renal Registry. Estimated life expectancy in a Scottish cohort with type 1 diabetes, 2008-2010. JAMA. 2015 Jan 6;313(1):37-44. doi: 10.1001/jama.2014.16425. PMID 25562264
- [Background] Rhodes ET, Prosser LA, Hoerger TJ, Lieu T, Ludwig DS, Laffel LM. Estimated morbidity and mortality in adolescents and young adults diagnosed with Type 2 diabetes mellitus. Diabet Med. 2012 Apr;29(4):453-63. doi: 10.1111/j.1464-5491.2011.03542.x. PMID 22150528
- [Background] Dabelea D, Stafford JM, Mayer-Davis EJ, D'Agostino R Jr, Dolan L, Imperatore G, Linder B, Lawrence JM, Marcovina SM, Mottl AK, Black MH, Pop-Busui R, Saydah S, Hamman RF, Pihoker C; SEARCH for Diabetes in Youth Research Group. Association of Type 1 Diabetes vs Type 2 Diabetes Diagnosed During Childhood and Adolescence With Complications During Teenage Years and Young Adulthood. JAMA. 2017 Feb 28;317(8):825-835. doi: 10.1001/jama.2017.0686. PMID 28245334
- [Background] Bryden KS, Peveler RC, Stein A, Neil A, Mayou RA, Dunger DB. Clinical and psychological course of diabetes from adolescence to young adulthood: a longitudinal cohort study. Diabetes Care. 2001 Sep;24(9):1536-40. doi: 10.2337/diacare.24.9.1536. PMID 11522695
- [Background] Bryden KS, Dunger DB, Mayou RA, Peveler RC, Neil HA. Poor prognosis of young adults with type 1 diabetes: a longitudinal study. Diabetes Care. 2003 Apr;26(4):1052-7. doi: 10.2337/diacare.26.4.1052. PMID 12663572
- [Background] Johnson B, Elliott J, Scott A, Heller S, Eiser C. Medical and psychological outcomes for young adults with Type 1 diabetes: no improvement despite recent advances in diabetes care. Diabet Med. 2014 Feb;31(2):227-31. doi: 10.1111/dme.12305. Epub 2013 Sep 19. PMID 23952498
- [Background] Rodwell L, Romaniuk H, Nilsen W, Carlin JB, Lee KJ, Patton GC. Adolescent mental health and behavioural predictors of being NEET: a prospective study of young adults not in employment, education, or training. Psychol Med. 2018 Apr;48(5):861-871. doi: 10.1017/S0033291717002434. Epub 2017 Sep 6. PMID 28874224
- [Background] 2014 Diabetes Health Care Cost Institute Utilization Report. Health Care Cost Institute. Published 2014. Accessed October 3, 2021. https://healthcostinstitute.org/images/easyblog_ articles/276/HCCI-2017-Health-Care-Cost-and-Utilization-Report-02.12.19.pdf
- [Background] Sequeira PA, Pyatak EA, Weigensberg MJ, Vigen CP, Wood JR, Ruelas V, Montoya L, Cohen M, Speer H, Clark S, Peters AL. Let's Empower and Prepare (LEAP): Evaluation of a Structured Transition Program for Young Adults With Type 1 Diabetes. Diabetes Care. 2015 Aug;38(8):1412-9. doi: 10.2337/dc14-2577. Epub 2015 Apr 23. PMID 25906787
- [Background] Pyatak EA, Carandang K, Vigen CLP, Blanchard J, Diaz J, Concha-Chavez A, Sequeira PA, Wood JR, Whittemore R, Spruijt-Metz D, Peters AL. Occupational Therapy Intervention Improves Glycemic Control and Quality of Life Among Young Adults With Diabetes: the Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) Randomized Controlled Trial. Diabetes Care. 2018 Apr;41(4):696-704. doi: 10.2337/dc17-1634. Epub 2018 Jan 19. PMID 29351961
- [Background] Bakhach M, Reid MW, Pyatak EA, Berget C, Cain C, Thomas JF, Klingensmith GJ, Raymond JK. Home Telemedicine (CoYoT1 Clinic): A Novel Approach to Improve Psychosocial Outcomes in Young Adults With Diabetes. Diabetes Educ. 2019 Aug;45(4):420-430. doi: 10.1177/0145721719858080. Epub 2019 Jun 27. PMID 31244396
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] American Diabetes Association 85th Scientific Sessions. Identifying Diabetes Distress across Adult Age Groups-Insights from the ReDUCe Study.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05000021/ICF_000.pdf